CLINICAL TRIAL: NCT04290273
Title: Characterisation of the Time-course Response of UV-induced Erythema
Acronym: CHERY
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: workforce issues which made practical delivery of the study impossible to do atthe current time
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government)
Responsible Party: Principal Investigator, Sally Ibbotson, Professor (Clinical), University of Dundee
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2-004-20
Record Dates: First submitted 2020-02-26; First posted 2020-02-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Erythema
Keywords: erythema; photobiology; photomedicine; phototherapy
MeSH Terms: conditions — Erythema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning exposure in week 1 (Experimental): Participants will have their first week of testing starting in the morning
  Interventions: Diagnostic Test: MED Test; Device: Wearing device
- Afternoon exposure in week 1 (Experimental): Participants will have their first week of testing starting in the afternoon
  Interventions: Diagnostic Test: MED Test; Device: Wearing device

INTERVENTIONS:
Diagnostic Test: MED Test — Participant is irradiated with several doses of UV light on small areas of the outer thigh. 24 hours later this area is visually inspected for erythema, and the minimal erythemal dose (MED) is determined.
Device: Wearing device — Participants wear a portable erythema measurement device for 48 hours. The device shines light on the skin at frequent intervals and measures skin 'redness'. The device is removed by a technician after the 48 hours.

SUMMARY:
Erythema is a physiological response to an insult on the skin. One such insult is ultraviolet (UV) radiation, with the resultant erythema also known as sunburn. It is a reddening of the skin as a result of increased blood flow to the area. By controlled exposure to UV radiation, a minimal erythema dose (MED) indicative of threshold erythemal sensitivity to the exposure waveband may be determined - this is determined visually by a trained clinician as the dose of light required to cause a just perceptible reddening of the skin. The MED of a specific patient on a specific skin site is an important measurement - it can allow for determination of initial dose in UV phototherapy, provides an indication of background levels of photosensitivity in diagnostic phototesting and may be influenced by exogenous factors, such as photoactive drugs.

The erythema response has been measured previously using non-invasive hand-held devices for a variety of UV exposures, including narrow-band (NB-)UVB, UVA and UVA1. Typically, the participant will be exposed in the morning (t = 0h) and have a reading taken immediately after. These readings are assessed visually by a trained clinician, or occasionally reflectance devices are used quantify erythema. The participant will then return at the end of the working day (t ~ 8h) for another reading, and again the next morning for another reading (t ~ 24h). This results in large gaps in the knowledge of erythemal response over time.

In this study the investigators aim to characterise the erythema response as a result of UV insult using a wearable erythema device to take continual measurements. This would allow us to more accurately determine the time point of peak erythema, which would inform and potentially change our current practice in reading MEDs. The investigators have previous experience of studies using reflectance devices to measure erythema time course at fixed intervals, however there are still gaps in the knowledge of the time course response of erythema.

There is no expected health benefit to participants in this study, however they may gain a better understanding of their responses to ultraviolet light MED testing. Controlled UV exposures are commonplace in our practice in the Photobiology Unit and it is not foreseen that there are any risks to participation in the study.

The primary objective in this study is to determine when the peak erythema index occurs in a healthy volunteer group. Success of this outcome will help fill in these gaps in the knowledge about the time course of erythema. The secondary objective is to determine if there is any difference in MED and/or peak erythema if the UV exposure is delivered in the morning vs. the afternoon. The outcomes of the research will be 20 sets (2 per participant) of continuous 48-hour erythema measurements.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers. No clinically significant abnormality identified by evaluation of medical history, in particular no evidence of photosensitivity
* Adult males and females, >18 years only
* Capable of giving informed consent
* Able to understand and adhere to protocol requirements
* Skin phototype I - III

Exclusion Criteria:

* Contact allergy to adhesives tapes
* Abnormal rash/pigmentation on thighs
* Unable to give informed consent
* Known to have a light sensitive disorder
* Pregnant, breastfeeding or planning to conceive
* Skin phototype IV - VI
* Lack of space on thighs for test procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Measure 2x 48 hour erythema time courses on each participant | 6 months

SECONDARY OUTCOMES:
Measure 2 MEDs (minimal erythemal doses) in each participant, at morning and afternoon exposures each | 6 months

REFERENCES:
- [Background] Dolotov LE, Sinichkin YP, Tuchin VV, Utz SR, Altshuler GB, Yaroslavsky IV. Design and evaluation of a novel portable erythema-melanin-meter. Lasers Surg Med. 2004;34(2):127-35. doi: 10.1002/lsm.10233. PMID 15004824
- [Background] Man I, McKinlay J, Dawe RS, Ferguson J, Ibbotson SH. An intraindividual comparative study of psoralen-UVA erythema induced by bath 8-methoxypsoralen and 4, 5', 8-trimethylpsoralen. J Am Acad Dermatol. 2003 Jul;49(1):59-64. doi: 10.1067/mjd.2003.419. PMID 12833009
- [Background] Man I, Dawe RS, Ferguson J, Ibbotson SH. An intraindividual study of the characteristics of erythema induced by bath and oral methoxsalen photochemotherapy and narrowband ultraviolet B. Photochem Photobiol. 2003 Jul;78(1):55-60. doi: 10.1562/0031-8655(2003)0782.0.co;2. PMID 12929749